CLINICAL TRIAL: NCT02195193
Title: Integrating Depression Care in Acute Coronary Syndromes Patients in Low Resource Hospitals in China
Brief Title: Integrating Depression Care in Acute Coronary Syndromes Care in China
Acronym: I-Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Peking University Sixth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: I-CARE; R01MH100332 (NIH)
Record Dates: First submitted 2014-07-15; First posted 2014-07-21 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Acute Coronary Syndromes; Depression
Keywords: Health Services Research; Acute Coronary Syndromes; Depression; Integrated care
MeSH Terms: conditions — Acute Coronary Syndrome; Depression | interventions — Delivery of Health Care, Integrated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (UC) (No Intervention): The standard interventions from Clinical Pathway for Acute Coronary Syndromes in China-Phase 3 (CPACS-3) study that are limited to in-patient ACS care (refer to "Usual Care" [UC]), will be implemented in the participating hospitals, and hence will be received by all patients in both intervention (IC) and control (UC) groups; standardized cardiovascular disease education also will be provided to all participants.CPACS-3 registration number is NCT01398228
- Intervention Care (IC) (Experimental): Besides of the UC, an nurse-coordinated integrated care model for Acute Coronary Syndromes(ACS) and depression will be delivered to intervention group, including ACS secondary prevention therapies at and after discharge, screening and treatment of depression during hospitalization and after discharge.
  Interventions: Other: Integrated care

INTERVENTIONS:
Other: Integrated care — an integrated care model for ACS and depression delivered by a collaborative team composed of cardiologists/internists and nurses in the same rural county hospital. The collaborative team will be able to provide medical services for the diagnosis and treatment at acute phase of ACS during hospitalization, ACS secondary prevention therapies at and after discharge, and screening and treatment of depression depressive symptom during hospitalization and after discharge. The core of the interventions includes: depressidepressive symptomon screening and classification, individual counseling and medical treatment of depression, group counseling and health education, and follow-up for ACS and depression treatments compliance, IT- system- assisting theassisted management and necessary referral.
  Arms: Intervention Care (IC)

SUMMARY:
The overall goal of this study is to develop, pilot test, implement, and evaluate a nurse-coordinated depression care model integrated into the care of Acute Coronary Syndromes (ACS) patients with rigorous assessment of feasibility, effectiveness, acceptability and cost in rural China. This study is a large multi-center, randomized clinical trial among 4,000 ACS patients from 20 rural county hospitals selected from a well-established research network across China.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 79 years old
* Hospitalized due to a diagnosis of Acute Coronary Syndromes (ACS)
* ACS is stable (as judged by the treating cardiologist/internist)
* Signed patient informed consent

Exclusion Criteria:

* Affected by severe cardiovascular disease or medical comorbidity that indicate the patient's life expectancy is less than 12 months (e.g. class IV heart failure, terminal cancer)
* Seriously disabled (unable to travel to the hospital, class IV heart failure at baseline)
* Suffering from problems that affect normal communication (e.g., intellectual impairment, observed mental confusion suggesting dementia, deafness, blindness, etc.)
* Non-permanent local residents or permanent residents planning to move out within 12 months
* Pregnant or breast-feeding or planning pregnancy within 12 months
* Affected by bipolar disorder, schizophrenia or severe depression that meet criteria for referral including patients with acutely suicidal risk (Beck Depression Inventory Item9=3)
* Having alcohol dependence (defined by MINI Alcohol Dependence/Abuse Part)

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4043 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Changes in mean Patient Health Questionnaire-9 (PHQ-9) score from baseline to 6 months | Before patient discharge and after 6 months from discharge
  Changes in mean Patient Health Questionnaire-9 (PHQ-9) score from baseline to 6 months
Changes in mean PHQ-9 score from baseline to 12 months | Before patient discharge and after 12 months from discharge
  Changes in mean Patient Health Questionnaire-9 (PHQ-9) score from baseline to 12 months

SECONDARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | At least 12 months after discharge
  MACE includes all cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, and re-hospitalization due to cardiovascular disease.
Proportion of patients with self-reported adherence to evidence-based Acute Coronary Syndromes (ACS) secondary prevention treatment at 6 and 12 months | At 6 and 12 months after discharge
  ACS secondary prevention treatment means combination use of aspirin, clopidogrel, statin, Angiotensin-Converting Enzyme Inhibitors/ Angiotensin Receptor Blocker and/or beta-blocker.
Quality of life (EQ5D) at 6 and 12 months after discharge | At 6 and 12 months after discharge

OTHER OUTCOMES:
Incidence of Major Adverse Events (MACE) after discharge | At 6 month and 12 month after patients discharged from hospital
  Includes all death, non-fatal myocardial infarction, non-fatal stroke, and re-hospitalization for any reasons after discharge
Proportion of patients with improved cardiovascular risk surrogates | At 6 month and 12 month after discharge
  Improved cardiovascular risk surrogates include blood pressure < 140/90 mmHg, heart rate < 70 beats/m, serum Low Density Lipoprotein-cholesterol < 100 mg/dL and blood sugar < 7.0 mmol/L
Proportion of patients with increased healthy life style | At 6 and 12 months after discharge
  Health life style includes physical activity >= 3 times/wk and more than 30 min. each time; no smoking, no alcohol use, and Body Mass Index (BMI) < 24 Kg/m2
Proportion of patients with self-reported adherence to general medicine treatment | At 6 and 12 months after discharge
  The Morisky scale has been used to measure patients' self-reported adherence
The interactions between the intervention effect on the outcomes and the modifiers | At 6 month or 12 month after discharge
  Modifiers include severity of depression measured by Patient Health Questionnaire-9(PHQ-9), events within or without 6 months after discharge, age and gender
Changes in mean Mini-International Neuropsychiatric Interview (MINI) score, Enriched social support instrument(ESSI) score and Perceived social support score (PSSS) score | Before patient discharge and at 6,12 months after discharge
  Subsample study. 800 patients from 4 hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Yangfeng Wu, MD, PhD, Principal Investigator — The Geogre Institute for Global Health, China
Locations (1):
- The George Institute for Global Health, China, Haidian, Beijing Municipality, China

REFERENCES:
- [Derived] Wu Y, Yu X, Zhu Y, Shi C, Li X, Jiang R, Niu S, Gao P, Li S, Yan L, Maulik PK, Guo G, Patel A, Gao R, Blumenthal JA. Integrating depression and acute coronary syndrome care in low resource hospitals in China: the I-CARE randomised clinical trial. Lancet Reg Health West Pac. 2024 Jul 1;48:101126. doi: 10.1016/j.lanwpc.2024.101126. eCollection 2024 Jul. PMID 39040037